CLINICAL TRIAL: NCT04737252
Title: Development and Initial Testing of a Couple-Based Intervention to Optimize Suicide and Self-Injury Treatment: COMPASS (Connecting, Overcoming, and Moving Past Suicide and Self-Injury)
Acronym: COMPASS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: York University (Other)
Collaborators: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Skye Fitzpatrick, Assistant Professor, York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG-0-057-19
Record Dates: First submitted 2020-12-17; First posted 2021-02-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Self-injurious Thoughts and Behaviours; Borderline Personality Disorder
Keywords: Self-injury Thoughts and Behaviours; Suicide; Non-suicidal Self-injury; Couple Intervention; Emotion Dysregulation; Intimate Relationship Dysfunction; Borderline Personality Disorder
MeSH Terms: conditions — Behavior; Borderline Personality Disorder; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Uncontrolled pilot trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sage (Experimental): Immediately receives 12 sessions of couple intervention aimed to improve self-injury thoughts and behaviours, emotion dysregulation, borderline personality disorder symptoms, and intimate relationship dysfunction.
  Interventions: Behavioral: Sage (formerly known as COMPASS)

INTERVENTIONS:
Behavioral: Sage (formerly known as COMPASS) — Sage is a remote 12 session intervention for couples wherein one individual has Borderline Personality Disorder (BPD) and engages in self-injury thoughts and behaviours. The intervention consists of elements of Cognitive Behavioural Conjoint Therapy (CBCT) and has been adapted for this population. Couples will meet remotely with a clinician (registered psychologists and/or graduate level clinicians) for 8-12 sessions via Zoom Healthcare. The primary outcomes are self-injury thoughts and behaviours (as measured by the Suicide Attempt and Self-Injury Interview-modified, and the Beck Scale for Suicidal Ideation and ecological momentary assessment) and borderline personality disorder symptoms (as measured by the Borderline Symptom List-23).

SUMMARY:
Self-injurious thoughts and behaviors (SITBs), including suicide, thinking about suicide, and self-injury without intent to die, are major public health crises, with variably effective, and sometimes long and expensive, interventions. SITBs are particularly common in borderline personality disorder (BPD). Moreover, people with BPD often cannot access SITB treatment, drop out of them, and may lose their improvements after them. Reducing SITBs in BPD requires innovative interventions that have greater impact and are faster to deliver. SITBs are particularly influenced by emotion dysregulation (i.e., intense, negative emotion and difficulties changing it) and intimate relationship dysfunction, but leading evidence-based SITB interventions typically focus on the former, while neglecting the latter. For other mental health problems, couple treatments result in comparable or better individual outcomes relative to individually-delivered treatments, with added benefits of enhanced intimate relationship functioning. SITB treatment outcomes in BPD could likely be expedited and optimized with a couple intervention that targets emotion dysregulation in a relational context and intimate relationship dysfunction. This project aims to develop, refine, and test a brief SITB intervention delivered conjointly to individuals with BPD and SITBs (i.e., "patients") and their intimate partners (i.e., "partners")- Sage (formerly known as COMPASS (Connecting, Overcoming, and Moving Past Suicide and Self- injury))- that targets both emotion dysregulation and intimate relationship dysfunction to reduce SITBs and BPD symptoms in the short- and long-term. Prior to formal testing in an uncontrolled trial, it is important to solicit preliminary data regarding the clarity, accessibility, safety, tolerability, and efficacy of Sage. This project involves 3 Phases: translating Sage outlines into a manual (Phase 1); refining Sage (Phase 2); and an uncontrolled pilot trial of Sage (Phase 3). In Phase 1, the three stages of Sage will be manualized to focus on (1) developing a conjoint safety plan to reduce SITB risk, (2) reducing emotion dysregulation and intimate relationship dysfunction, and (3) changing patterns that maintain SITBs. In Phase 2, Sage will be delivered to 5-10 patients with BPD and SITBs and their partners (i.e., 5-10 couples) who will provide feedback about whether Sage is clear, helpful, and useable. This feedback will be used to refine the Sage manual. In Phase 3, the investigators will test whether Sage is safe, initially efficacious, and feasible by administering it to 15-20 patients with BPD and SITB and their partners (i.e., 15-20 couples). The investigators will examine whether Sage results in changes in SITBs and BPD symptoms in patients with BPD and SITBs, and SITB risk factors (e.g., emotion dysregulation and intimate relationship dysfunction) in both patients and partners. These outcomes will be measured multiple times per day during treatment using participant's smartphones (i.e., ecological momentary assessment), and interviews/questionnaires administered at the beginning, middle, end, and at 3 months after the intervention. The investigators predict that Sage will reduce SITBs and BPD symptoms in the patient with BPD and SITBs and improve emotion dysregulation and intimate relationship dysfunction in both patients with BPD and SITBs and their partners. This study offers a novel SITB and BPD treatment that directly targets SITBs, BPD symptoms, and the factors that drive them. Its short duration broadens the accessibility of BPD and SITB interventions with the potential to contribute to reducing SITBs and BPD symptoms on a large scale. During this period of social distancing due to COVID-19, Sage will be delivered remotely via secure videoconferencing (Zoom Healthcare). As social distancing restrictions lift, Sage will be delivered in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have either engaged in 2+ suicidal or non-suicidal self-injurious behaviors in the past two weeks (i.e., chronic and recent SITBs, consistent with previous research evaluating non-suicidal self-injury (Kranzler et al., 2018)), or have severe suicidal ideation as indicated by a score ≥15 on the Beck Scale for Suicidal Ideation (Beck, 1991)
2. Patients also meet diagnostic criteria for BPD
3. Patients are between the ages of 18 and 70 years-old
4. Patients have a romantic partner who is between the ages of 18 and 70 years-old
5. Patient's romantic partner is willing to participate in the study with them

Exclusion Criteria:

1. Past-year severe intimate aggression in their relationship such that participants who endorse any severe physical and/or sexual assault behaviors in the past year will be excluded from the study (Monson et al., 2012; Abramowitz et al., 2013), as assessed by the Revised Conflict Tactics Scale, Severe Items Subscale (CTS-2; Straus, Hamby, Boney-McCoy, & Sugarman, 1996)
2. Either partner has a severe substance use disorder that would interfere with the capacity to attend and participate in this study
3. Either partner has clinically significant psychotic symptoms or bipolar I disorder (e.g., McMain et al., 2018; McMain et al., 2009)
4. Either partner has a major cognitive or intellectual impairment that would prevent the individual's ability to attend intervention and participate in the research study
5. Either partner has illiteracy in English language
6. Either partner is unable or unwilling to download and use a mobile application on their smart phone to complete daily Ecological Momentary Assessment (EMA) measures
7. If partners meet inclusion criterion #1, or #2, or meet the self-harm/suicidal behaviour diagnostic criterion for BPD.
8. If either partner of the couple is unwilling to have assessments and sessions audio or videorecorded
9. If either partner is currently not residing in Ontario

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the frequency and intensity of self-injury thoughts and behaviours from baseline will be examined through ecological momentary assessment. | It will be administered daily (three times per day) for five weeks throughout the intervention; from baseline to post intervention
Change in frequency of self-injury thoughts and behaviours from baseline, as measured by the Suicide Attempt Self-Injury Interview-modified. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
Change in severity of suicidal ideation from baseline, as measured by the Beck Scale for Suicidal Ideation. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Beck Scale for Suicidal Ideation has a minimum possible score of 0, and maximum possible score of 38, wherein higher scores reflect more severe suicidal ideation.
Changes in Borderline Personality Symptom severity from baseline, as measured by the Borderline Symptom List-23. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Borderline Symptom List-23 has a minimum possible score of 0, and maximum possible score of 92, wherein higher scores reflect more severe borderline personality disorder symptoms.
Changes in Borderline Personality Symptom severity from baseline, as measured by the Zanarini Rating Scale for Borderline Personality Disorder (self-report) | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Zanarini Rating Scale for Borderline Personality Disorder (self-report) has a minimum possible score of 0, and maximum possible score of 36, wherein higher scores reflect more severe borderline personality disorder symptoms.

SECONDARY OUTCOMES:
Change in severity of depression from baseline, as measured by the Patient Health Questionnaire-9. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Patient Health Questionnaire-9 has a minimum possible score of 0 and a maximum possible score of 27, wherein higher scores reflect higher severity of depression.
Changes is emotion dysregulation from baseline, as measured by The Difficulties in Emotion Regulation Scale (DERS). | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Difficulties in Emotion Regulation scale has a minimum possible score of 36, and maximum possible score of 180, wherein higher scores reflect greater emotion dysregulation.
Changes in one's report of their partner's emotion dysregulation from baseline, as measured by the Difficulties in Emotion Regulation Scale - Partner Version (DERS-Partner). | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Difficulties in Emotion Regulation Scale - Partner has a minimum possible score of 8, and maximum possible score of 40, wherein higher scores reflect more severe emotion dysregulation reported of one's partner.
Changes in severity of conflict from baseline, as measured by the Ineffective Arguing Inventory. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Ineffective Arguing Inventory has a minimum possible score of 8, and a maximum possible score of 40, wherein higher scores indicate decreased satisfaction with the style of arguing in a relationship.

OTHER OUTCOMES:
Changes in participants psychiatric and medical treatments (e.g., medication, day treatment programs) from baseline, measured by The Mental Health Utilization Interview-Modified. | It will be administered only at baseline (pre-intervention) and immediately after the intervention.
Changes in relationship satisfaction from baseline, as measured by mean change from baseline on the Couples Satisfaction Index. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Couples Satisfaction Index has a minimum possible score of 0, and a maximum possible score of 161, wherein higher scores reflect higher levels of relationship satisfaction.
Changes in severity of Anxiety from baseline, as measured by Generalized Anxiety Disorder-7. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Generalized Anxiety Disorder-7 has a minimum possible score of 0 and maximum possible score of 21, wherein higher scores reflect more severe levels of anxiety.
Changes in Posttraumatic Stress Disorder severity from baseline, as measured by the Post-Traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). | It will be administered only half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Post-Traumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) has a minimum possible score of 0 and a maximum possible score of 80, wherein higher scores reflect more severe posttraumatic stress disorder symptomatology.
Changes in one's report of their partner's Borderline Personality Symptoms severity from baseline, as measured by the Borderline Symptom List-23 - Partner Report. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
Changes in suicidal ideation severity from baseline, as measured by the Suicide Behaviours Questionnaire-Revised. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Suicide Behaviours Questionnaire-Revised has a minimum possible score of 3, and a maximum possible score of 18, wherein higher scores indicate more severe suicidal ideation.
Changes in one's report of their partner's suicidal ideation from baseline, as measured by the suicide Behaviours Questionnaire-Revised - Partner Report. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Suicide Behaviours Questionnaire-Revised - Partner Report has a minimum possible score of 3, and a maximum possible score of 18, wherein higher scores indicate more severe suicidal ideation reported of their partner.
Changes in emotional reactivity from baseline, as measured by the Emotional Reactivity. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Emotional Reactivity Scale has a minimum possible score of 0, and a maximum possible score of 84, wherein higher scores reflect greater emotional reactivity.
Changes in affect from baseline, as measured by the Positive and Negative Affect Schedule-Modified. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
Changes in addiction severity from baseline, as measured by the Addiction Severity Index. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
Changes in Work, Health, and Life Quality from baseline, as measured by 3 one-item self-report measurements that assess work functioning, perceived health status, and overall quality of life. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
Changes in shame from baseline, as measured by the Experience of Shame Scale. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
  The Experience of Shame Scale has a minimum possible score of 25, and a maximum possible score of 100, wherein higher scores reflect higher levels of shame.
Frequency of Emergency Department Visits and Hospitalizations with change measured as mean change from baseline. | It will be administered only at baseline (pre-intervention), half-way through intervention, immediately after the intervention, and three months after the intervention (Phase 3 only).
Client satisfaction with the intervention as measured by the Client Satisfaction Questionnaire. | It will be administered only immediately after the intervention
  The Client Satisfaction Questionnaire has a minimum possible score of 8, and a maximum possible score of 32, wherein higher scores reflect greater satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Skye Fitzpatrick, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzpatrick S, Wagner AC, Monson CM. Optimizing borderline personality disorder treatment by incorporating significant others: A review and synthesis. Personal Disord. 2019 Jul;10(4):297-308. doi: 10.1037/per0000328. Epub 2019 Feb 4. PMID 30714800
- [Background] Fitzpatrick S, Liebman RE, Monson CM. The borderline interpersonal-affective systems (BIAS) model: Extending understanding of the interpersonal context of borderline personality disorder. Clin Psychol Rev. 2021 Mar;84:101983. doi: 10.1016/j.cpr.2021.101983. Epub 2021 Jan 24. PMID 33517245
- [Derived] Fitzpatrick S, Varma S, Traynor J, Earle EA, Vanstone R, Fulham L, Goenka K, Blumberg MJ, Wyatt L, Siegel AN, Di Bartolomeo AA, Norouzian N, Burdo J, Ennis N, Carney A, Luxor O, Sankar R, Monson C, Liebman R. A pilot and feasibility study of Sage: A couple therapy for borderline personality disorder. Psychother Res. 2025 Apr 15:1-16. doi: 10.1080/10503307.2025.2491478. Online ahead of print. PMID 40233277
- [Derived] Fitzpatrick S, Varma S, Chafe D, Norouzian N, Traynor J, Goss S, Earle E, Di Bartolomeo A, Siegel A, Fulham L, Monson CM, Liebman RE. A case series of sage: a new couple-based intervention for borderline personality disorder. Borderline Personal Disord Emot Dysregul. 2024 Jan 12;11(1):1. doi: 10.1186/s40479-023-00244-x. PMID 38212804